CLINICAL TRIAL: NCT05202522
Title: Dancing to Improve Mobility and Cognition: A Feasibility Randomized Control Trial of Virtual GERAS DANCE
Brief Title: Virtual GERAS DANCE Feasibility RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 14400
Record Dates: First submitted 2022-01-07; First posted 2022-01-21 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2022-03

CONDITIONS: Aging
Keywords: Dance; Exercise; Rehabilitation
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): During the study. participants in the control group will not receive the virtual GERAS DANCE intervention. However, they will receive the virtual GERAS DANCE intervention following study completion for equal opportunity to participate in the program.
- Virtual GERAS DANCE Group (Experimental): Virtual GERAS DANCE will be delivered for 1-hr twice weekly for 6 weeks.
  Interventions: Behavioral: Virtual GERAS DANCE

INTERVENTIONS:
Behavioral: Virtual GERAS DANCE — Dance is a form of aerobic exercise that involves multicomponent training with physical, cognitive, and social dimensions and may have synergetic benefits when delivered in combination. GERAS DANcing for Cognition and Exercise (DANCE), a community-based rehabilitation program for older adults with cognitive decline and/or mobility impairments, has been adapted for virtual delivery through videoconferencing systems. Participants will receive twice-weekly (one hour per session) virtual dance sessions for a total of 6 weeks.
  Arms: Virtual GERAS DANCE Group

SUMMARY:
GERAS DANcing for Cognition and Exercise (DANCE) is a therapeutic mind-body program for older adults (aged 60+) developed with rehabilitation and geriatric medicine expertise at the GERAS Centre for Aging Research at Hamilton Health Sciences and McMaster University. This study will examine if a virtual dance program is feasible for older adults and if dancing at home can benefit mind-body health, self-confidence, and mood.

DETAILED DESCRIPTION:
GERAS DANCE fulfills an urgent need in our community to provide tailored evidence-based programming to help improve the health of older adults and was adapted for virtual implementation. This randomized controlled trial (RCT) aims to measure (1) the feasibility of virtual GERAS DANCE in older adults to inform a large full-scale study, and (2) the potential effects of virtual GERAS DANCE on mobility, balance self-efficacy, cognition, frailty, and mood in older adults. This study will utilize a single-center, prospective, parallel-group randomized controlled feasibility approach. This RCT will involve 48 older adults using a person-centered and coordinated model of care embedded into existing community health partnerships. Participants will be randomized to receive 6-weeks of virtual GERAS DANCE or usual care. All participants randomized to usual care will receive the dance intervention after study completion for equal opportunity to participate in the virtual GERAS DANCE program. The progressive GERAS DANCE curricula will be delivered virtually for 1-hr class twice weekly by a certified GERAS DANCE instructor. GERAS DANCE curricula include gradual increases in cognitive load and are based on motor learning principles of the ABCs of movement Agility, Balance, and Coordination. The ABCs of movement is essential to quickly and efficiently change the body position with balance and coordination. Assessments of mobility, balance self-efficacy, cognition, frailty, and mood will occur at baseline and 6-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling adults aged ≥ 60 years of age;
* Has access, or has a caregiver who has access to a device at home that can support a videoconferencing service
* Able to ambulate independently with or without a walking aid; OR with caregiver supervision at home;
* Family physician's signature on a medical clearance form to ensure they are cleared to exercise safely.

Exclusion Criteria:

* Unable to speak or understand English and has no caregiver for translation;
* Significant cognitive impairment where they may have difficulty following two-step commands;
* Unstable angina or unstable heart failure;
* Travel plans that would result in missing greater than 20% of the trial's 6-week duration;
* Currently attending a group exercise program.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | [Time Frame: Through study completion, an average of 10 months]
  5 patient/month
Retention Rate | [Time Frame: Through study completion, an average of 10 months]
  target ≥ 70%
Data Collection completion | [Time Frame: Through study completion, an average of 10 months]
  target ≥ 70%
Proportion of recruited patients | [Time Frame: Through study completion, an average of 10 months]
  target ≥ 70%
Refusal Rate | [Time Frame: Baseline, 6-weeks]
  target ≥ 70%

SECONDARY OUTCOMES:
Change in Mobility | Baseline and 6 Weeks
  Assessed by the 5x Sit-to-Stand (time to complete). Faster times to complete indicate better performance.
Change in Balance | Baseline and 6 Weeks
  Balance confidence will be assessed using the Activities-specific Balance Confidence Scale (ABCs). Higher scores indicate greater balance confidence [range 0-100].
Change in Falls Self-Efficacy | Baseline and 6 Weeks
  Level of concern for falling will be assessed using the Falls Efficacy Scale - International (FES-I). Higher scores indicate greater concern for falling [range 1-4].
Change in Frailty | Baseline and 6 Weeks
  Assessed by Fit-Frailty App. Higher scores indicate greater degree of frailty [range 0-1].
Change in Cognition | Baseline and 6 Weeks
  Assessed by Telephone-based Montreal Cognitive Assessment (MoCA). Higher scores indicate better cognition [range 0-30].
Change in Mood | Baseline and 6 Weeks
  Assessed by Depression Anxiety Stress Scale (DASS-21) Questionnaire. Higher scores indicate greater depression [range 0-120].

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Papaioannou, MD, MSc, Principal Investigator — Scientific Director, GERAS Centre for Aging Research
Locations (1):
- McMaster University - St. Peter's Hospital, Hamilton, Ontario, Canada